CLINICAL TRIAL: NCT02369627
Title: Facilitating HIV Testing Among Young Adult MSM Through Social Networking
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Roland C. Merchant, MD. MPH, ScD, Associate Professor of Emergency Medicine and Epidemiology at Alpert Medical School of Brown University and Rhode Island Hospital, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 477192-10
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: HIV
MeSH Terms: interventions — Residence Characteristics

ARMS (3):
- Rapid HIV Self-Test (Experimental): Participants will perform a rapid HIV self-test using the OraQuick® In-home HIV Test.
  Interventions: Device: Rapid HIV Self-Test (OraQuick® In-home HIV Test)
- Conventional Home-Based HIV Test (Active Comparator): Participants will perform a conventional home-based HIV test using the Home Access Express HIV-1 Test System.
  Interventions: Device: Conventional Home-Based HIV Test (Home Access Express)
- Community/Medical-Based HIV Test (Active Comparator): Participants will receive a link to a CDC website (https://gettested.cdc.gov) that allows them to search for HIV testing locations of their choice.
  Interventions: Other: Community/Medical-Based HIV Test

INTERVENTIONS:
Device: Rapid HIV Self-Test (OraQuick® In-home HIV Test) — The participant will utilize materials and directions contained within the OraQuick In-Home HIV Test kit to properly perform a rapid HIV self-test. The participant will first swab his upper and lower gums using an Oral Swab Test Stick. The participant will then place this device in a test tube, and the results will be displayed in the Test Window within 20 minutes. Test results expire after 40 minutes.
  Arms: Rapid HIV Self-Test
Device: Conventional Home-Based HIV Test (Home Access Express) — The participant will utilize materials and directions contained within the Home Access Express HIV-1 Test System to properly perform a conventional home-based HIV test. The participant is required to gather a blood sample by lancing his finger. Blood samples are collected by placing drops of blood on a packaged specimen card. The participant will then mail his blood sample to the Home Access laboratory using a self-addressed, pre-paid shipping envelope. The Home Access laboratory will process the blood sample, and the participant is required to call the facility to learn his HIV test result.
  Arms: Conventional Home-Based HIV Test
Other: Community/Medical-Based HIV Test — The participant will receive a link to a CDC website (https://gettested.cdc.gov) to search for HIV testing locations in his surroudning community. This resource website will provide the participant with places that offer HIV testing for free or at a low cost. The participant also has the option of going to places that can use his insurance or charge for testing. The pariticant is responsible to pay for any testing costs.
  Arms: Community/Medical-Based HIV Test

SUMMARY:
The purpose of this study is to evaluate a new approach to increase HIV testing among young adult Black, Hispanic, and white men-who-have-sex-with-men (MSM). In this randomized, controlled trial, participants will be assigned to one of three HIV testing groups: (1) rapid HIV self-testing group (OraQuick® In-home HIV Test), (2) conventional "home-based" HIV testing group (Home Access Express), and (3) community/medical-based HIV testing group. Upon completion of testing, participants will receive a questionnaire to evaluate their HIV testing experience, and also inquire about recommendations for future testing. Study participants will also have the option to refer other study eligible males to the study via email.

DETAILED DESCRIPTION:
Young adult (18-24-year-old) Black, Hispanic, and white men-who-have-sex-with-men (MSM) have among the highest incidences of new HIV infections in the US yet have low HIV testing rates. Access, cost, time, and concerns about confidentiality are some of the barriers that limit these men from being tested at traditional medical/community-based testing sites. A new US Food and Drug Administration-approved rapid HIV self-test (OraQuick® In-home HIV Test) might encourage and facilitate HIV testing because of its widespread access, convenience, ease of usage, oral fluid collection system, privacy, and rapid provision of test results. Despite these advantages, the investigators do not know if the new rapid HIV self-test will be preferred over medical/community-based or conventional "home-based" HIV testing, and if it will serve as a means of improving HIV testing use among young adult MSM.

The objectives of this study are to: (1) determine if testing uptake is higher in a rapid HIV self-testing group than in a conventional "home-based" HIV testing group and a community/medical-based testing referral group; (2) determine if time to initiation of HIV testing is shorter in the rapid HIV self-testing group, as compared to the other two participant groups; (3) determine if participants are more willing to contact and refer other young adult MSM to this study to use a rapid HIV self-test vs. a conventional "home-based" HIV test, or vs. a community/medical-based HIV test; (4) determine if those referred for rapid HIV self-testing are more likely to enroll in the study, have a higher uptake of testing, and have a shorter time to initiate HIV testing than those referred for conventional "home-based" HIV test, or a community/medical-based HIV test.

This study is comprised of three stages, the first of which is closed. In Stage I of this study, the investigators surveyed a large sample of MSM social-networking website users and assessed their acceptance, facilitators/barriers to use, utilization, preferences, and opinions regarding the new rapid HIV self-test, as compared to conventional "home-based" HIV testing or medical or community-based HIV testing. Of the participants enrolled in Stage I, 150 Black, 150 Hispanic, and 150 white MSM will be invited to participant in Stage II of this study. In this randomized, controlled trial, participants will be assigned to one of three HIV testing groups: (1) rapid HIV self-testing group (OraQuick® In-home HIV Test), (2) conventional "home-based" HIV testing group (Home Access Express), and (3) community/medical-based HIV testing group. Participants assigned to the rapid and conventional HIV testing groups will receive an internet-based coupon to order a free HIV testing kit from a specified pharmacy's website that will be delivered to the address of their choosing. The rapid HIV self-test kit and the conventional "home-based" HIV test kit contain all materials and instructions needed to conduct an HIV test. Participants assigned to the community/medical-based HIV testing group will receive a link to a CDC website (https://gettested.cdc.gov) that allows them to search for HIV testing locations of their choice. Participants in all three groups will receive an email explaining that the investigators are measuring uptake and time to testing among study participants. They will also be informed that the investigators will contact them after they have been tested to ask for their opinions regarding their testing experience. At the end of Stage II, participants will have the opportunity to refer other young adult MSM to the study via email. Referral participants will encompass Stage III of the study. Stage III participants will be assigned to the same testing group as the individual who referred them. Confidentiality will be maintained throughout all three stages of this study.

ELIGIBILITY:
Inclusion Criteria:

* Stage II inclusion criteria is contingent upon the enrollment and completion of Stage I of this study.
* Stage III inclusion criteria include: (1) 18-24 year-old male; (2) US resident; (3) previously had anal intercourse (insertive or receptive) with at least one male partner; (4) known to be HIV negative.

Exclusion Criteria:

* Female

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 425 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02-28 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Facilitating HIV Testing Among Young Adult MSM Through Social Networking Questionnaire | Three Months

CONTACTS AND LOCATIONS:
Overall Officials: Roland C Merchant, MD, Principal Investigator — Rhode Island Hospital

REFERENCES:
- [Derived] Wentz AE, Merchant RC, Clark MA, Liu T, Rosenberger JG, Bauermeister JA, Mayer KH. Blood Donation, Sexual Practices, and Self-Perceived Risk for HIV in the United States Among Young Adult Men Who Have Sex With Men. Public Health Rep. 2019 Jan/Feb;134(1):36-46. doi: 10.1177/0033354918815182. Epub 2018 Dec 7. PMID 30526313
- [Derived] Merchant RC, Clark MA, Liu T, Romanoff J, Rosenberger JG, Bauermeister J, Mayer KH. Comparison of Home-Based Oral Fluid Rapid HIV Self-Testing Versus Mail-in Blood Sample Collection or Medical/Community HIV Testing By Young Adult Black, Hispanic, and White MSM: Results from a Randomized Trial. AIDS Behav. 2018 Jan;22(1):337-346. doi: 10.1007/s10461-017-1802-x. PMID 28540562